CLINICAL TRIAL: NCT02458430
Title: Cholinergic Mechanisms of Gait Dysfunction in Parkinson's Disease - Clin Core/Proj#2
Brief Title: Cholinergic Mechanisms of Gait Dysfunction in Parkinson's Disease
Acronym: UDALL
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Principal Investigator, University of Michigan
Other Study IDs: HUM00093414
Record Dates: First submitted 2015-03-18; First posted 2015-06-01 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Balance and gait problems cause severe impairments for people with Parkinson's disease In some Parkinson's disease patients the investigators see a loss of acetylcholine in the brain. In previous studies the investigators have shown that this loss of acetylcholine is related to impaired balance and gait function in Parkinson's disease. In this study the investigators will take a closer look at this finding.

DETAILED DESCRIPTION:
Balance and gait problems cause severe impairments for people with Parkinson's disease and significantly affect their quality of life. Several changes occur in the brains of Parkinson's disease patients. The hallmark change is a loss of a neurotransmitter ("chemical messenger" between brain cells) called dopamine. To alleviate Parkinson's disease symptoms doctors prescribe dopamine replacement therapy, for example Sinemet (levodopa). Although effective for some of the symptoms, it typically does not sufficiently alleviate balance and gait problems. This study focuses on other changes in the brain that occur in Parkinson's disease that may contribute to balance and gait problems. In particular we will be looking at another neurotransmitter called acetylcholine. In some Parkinson's disease patients we see a loss of acetylcholine in the brain. In previous studies we have shown that this loss of acetylcholine is related to impaired balance and gait function in Parkinson's disease. In this study we will take a closer look at this finding.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and above (M/F).
2. PD diagnosis (with or without mild cognitive impairment; MCI) will follow the UK Parkinson's Disease Society Brain Bank Research Center (UKPDSBRC) clinical diagnostic criteria for PD (47), consistent with the typical nigrostriatal denervation pattern on VMAT2. Absence of significant dementia confirmed by neuropsychological testing. Modified Hoehn and Yahr stages 1-4 (48, 49).
3. PSP diagnosis will follow the NINDS-PSP clinical diagnostic criteria (50, 51).
4. All PD subjects will be required to have nigrostriatal dopaminergic denervation as demonstrated by [11C]DTBZ PET imaging (52, 53). Subjects with Parkinsonism and absence of this PD-typical pattern will be re-categorized .

Exclusion Criteria:

* 1. Presence of significant dementia. 2. Disorders which may resemble PD or PSP, such as dementia with Lewy bodies, vascular dementia, normal pressure hydrocephalus, multiple system atrophy, corticobasal ganglionic degeneration, or toxic causes of parkinsonism. The use of the UKPDSBRC and NINDS-PSP clinical diagnostic criteria will mitigate the inclusion of patients with atypical parkinsonism.

  3. Subjects on neuroleptic (except for low dose quetiapine 25-50 mg/d), anticholinergic (trihexyphenidyl, benztropine), cholinesterase inhibitors. Subjects with prior exposure to disallowed medications may be eligible if there has been an interval of > 2 months off these medications.

  4. Evidence of a large vessel stroke in a clinically relevant area (cerebral cortex, basal ganglia, thalamus) or mass lesion on structural brain imaging (MRI or CT).

  5. Participants in whom magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.

  6. Severe claustrophobia precluding MR or PET imaging. 7. Subjects limited by previous participation in research procedures involving ionizing radiation.

  8. Pregnancy (test within 48 hours of each PET session) or breastfeeding 9. History of deep brain stimulation surgery.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ago 50 and over
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-01-05; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
to assess change in balance and gait | data/testing is obtained at the initial visit and at a 2 year year follow up to note any changes in balance and gait
  motor tests are administered in an "off" state (by delaying the time at which the subject takes prescribed medication, subjects take their prescribed PD meds after the test battery, then tests are repeated one hour later in an "on" state. This is done at the initial study visit and at the 2 year follow up visit
to assess change in memory and cognition | data/testing obtained at the initial visit and at a 2 year follow up to note any changes for memory and cognition
  the same test battery of neuropsychology tests is administered at the initial study visit and at the 2 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, MD PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System Functional Neuroimaging, Cognitive and Mobility Laboratory, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Barr J, Vangel R, Kanel P, Roytman S, Pongmala C, Albin RL, Scott PJH, Bohnen NI. Topography of Cholinergic Nerve Terminal Vulnerability and Balance Self-Efficacy in Parkinson's Disease. J Integr Neurosci. 2024 Sep 24;23(9):178. doi: 10.31083/j.jin2309178. PMID 39344233